CLINICAL TRIAL: NCT06105372
Title: Effects of Ramadan Fasting on the Intestinal Microbiota and Fatty Acid Binding Protein 4 (FABP4) of Individuals
Brief Title: Ramadan Fasting, Microbiota and FABP4
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Aylin Seylam Küşümler, Assistant Professor, Okan University
Other Study IDs: 1969
Record Dates: First submitted 2023-10-13; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Intermittent Fasting
Keywords: Fasting, Microbiota; Fatty Acid-Binding Proteins
MeSH Terms: conditions — Intermittent Fasting; Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study, which aims to examine the effect of Ramadan fasting on intestinal microbiota composition and FABP4, was designed as a quasi-experimental study.

This study is planned to be conducted with volunteer participants who fasted during the Ramadan and met the inclusion criteria.

DETAILED DESCRIPTION:
The sample of the study was determined as 10 volunteer male participants who fasted during the Ramadan and met the inclusion criteria. Participants will not be subjected to any energy restriction, they will be fed ad-libitum and only the effect of intermittent fasting and fasting time on the variables will be examined.

Intermittent fasting is supported by increasing studies showing that it has a purifying effect on health. In particular, fasting practices exceeding 16 hours induce autophagy at the cellular level and this continues its effect in all tissue and organ systems after the regeneration movement that starts at the cellular level.

One of the important factors affected by intermittent fasting is the changes in microbiota, which is closely related to the general health of humans. Microbiota is generally defined as the colonization of certain places in our body by various populations of microorganisms and is affected by many factors such as nutrition, lifestyle, exercise, drug use and stress.

Fatty acid binding protein 4 (FABP4) is an adipocyte member of the fatty acid binding protein (FABP) family with nine different isoforms. It is highly secreted from adipose tissue but is also expressed from monocytes, macrophages and dendritic cells. This adipocyte, which increases in obesity, is found at higher levels in women than in men. Studies have shown that increased serum FABP4 levels are associated with Type 1 and Type 2 diabetes mellitus (DM), insulin resistance, and cardiovascular diseases.

The aim of this thesis study was to investigate the effect of Ramadan fasting on gut microbiota and FABP4.

The hypotheses of the study were;

1. Gut microbiota composition of adult individuals differs before and after Ramadan fasting.
2. Serum FABP4 and other biochemical values of adult individuals differ before and after Ramadan fasting.
3. Anthropometric measurements of adults differ before and after Ramadan fasting. All individuals who meet the inclusion and exclusion criteria and agree to participate in the study will be read and signed the Informed Voluntary Consent Form and a copy will be delivered to them. Questions related to the socio-demographic status and dietary habits of all participants will be asked to them and recorded in the questionnaire form by the researcher using the face-to-face interview technique.

Information about the volunteers who participated in the study, such as not having any disease (DM, hypertension, dyslipidemia, cancer, chronic renal failure, GI problems, etc.), not taking medication, and not having used antibiotics in the last six months, were evaluated by the Specialist Dr. who took part in the study. Dr. evaluated the participants through a preliminary interview with the participants. Factors such as the fact that the volunteers who participated in the study did not drink alcohol, had not applied for any diet program in the last six months, whether the participants were doing sahur or not, and especially that all participants had the same duration of fasting during the day during Ramadan were evaluated by the researcher through a preliminary interview with the participants. All individuals who met the inclusion and exclusion criteria and agreed to participate in the study were read and signed the Informed Voluntary Consent Form and a copy was delivered to them.

In order to evaluate the nutritional status of the individuals, the participants will be asked to record the amount of food consumption one week before the start of Ramadan fasting and during the last week of Ramadan for three consecutive days, one day of which will coincide with the weekend, and what should be considered during recording will be explained with examples in advance.

A physical activity record form will be filled out to determine the 24-hour physical activity status of the individuals included in the study and daily energy expenditure will be calculated.

With the start of the study, all participants will be asked about their food consumption records for 3 days (2 days on weekdays + 1 day on weekends), anthropometric measurements (body weight, height, waist circumference, hip circumference) and 24-hour physical activity records one week before the start of Ramadan fasting and the last week of Ramadan.

One day before and on the last day of Ramadan fasting, fecal and blood samples will be collected and total microbiota, FABP4, CRP, fasting insulin, fasting blood glucose, HDL-C, LDL-C, Total-C, TG, ALT, AST and GGT values will be analyzed and recorded.

Descriptive statistics will be given as number and percentage for categorical variables and arithmetic mean and standard deviation for continuous variables. Chi-square test will be used to compare categorical variables. Whether the research data are suitable for normal distribution or not will be tested with Kolmogorov-Smirnov analysis method, and when parametric test assumptions are met in the comparison of independent group differences, t test and Analysis of Variance will be used in independent groups; Mann-Whitney U test and Kruskal Wallis tests will be used when parametric test assumptions are not met. In the comparison of dependent groups, if parametric assumptions are met, t test and repeated measures analysis of variance will be used; Wilcoxon test and Friedman test will be used when parametric test assumptions are not met. Statistical significance level p<0.05 will be accepted.

ELIGIBILITY:
Inclusion Criteria:

1. Not having a chronic disease diagnosed by a doctor (DM, hypertension, dyslipidemia, cancer, chronic renal failure, GI problems, etc.)
2. Being a male between the ages of 20-50
3. Body mass index (BMI) > 18.5 and < 34.9 kg/m2
4. Not drinking alcohol
5. Not having applied any diet program in the last 6 months
6. Not taking prebiotic or probiotic supplements in the last 6 months
7. Not having used antibiotics in the last 6 months
8. Not using nutritional supplements
9. Volunteering to participate in the research

Exclusion Criteria:

* Women will not be included in the study due to the fact that they will not be able to fast the entire Ramadan fast due to menstruation.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample of the study was determined as 10 volunteer male participants who fasted during the Ramadan and met the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
BMI (kg/cm2) | Pre-procedure, after 4 weeks
  After measuring the body weight (kg) and height (m) of the individuals participating in the study, BMI (kg/m2) values will be calculated; weight and height will be combined to report BMI in kg/m^2 according to the formula [body weight (kg) / height2 (m2)].
Physical activity levels | Pre-procedure, after 4 weeks
  In the calculation of physical activity levels, the equation [(Physical activity rate (PAR) for Activity Type x Duration of Activity (hours)) / (total duration (1440)] will be used.
Food consumption record | one week before the procedure and up to 4 weeks
  Record food consumption for three consecutive days, with one day falling on a weekend
Microbiota analysis | Pre-procedure, after 4 weeks
  Fecal will be collected from participants and total microbiota will be analyzed.
FABP4 analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and FABP4 (ng/L) values will be analyzed and recorded.
CRP analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and CRP(mg/L) will be analyzed and recorded.
HDL-C analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and HDL-C (md/dl) will be analyzed and recorded.
LDL-C analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and LDL-C (md/dl) will be analyzed and recorded.
Total-C analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and Total-C (mg/dl) will be analyzed and recorded.
Tg analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and Tg (mg/dl) will be analyzed and recorded.
ALT analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and ALT (U/L) will be analyzed and recorded.
AST analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and AST (U/L) will be analyzed and recorded.
GGT analysis | Pre-procedure, after 4 weeks
  Blood samples will be collected from participants and GGT (U/L) will be analyzed and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- OkanU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No